CLINICAL TRIAL: NCT01855282
Title: Pasos Saludables: A Pilot Intervention to Prevent Obesity and Diabetes Among Latino Farm Workers
Brief Title: Assessment of an Intervention to Prevent Obesity and Diabetes in Latino Farm Workers
Acronym: Pasos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 219631; S-MSPREIT (Other: UC Davis)
Record Dates: First submitted 2013-05-08; First posted 2013-05-16 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Overweight and Obesity
Keywords: Diabetes Type II,; Overweight,; Obesity,; Behavioral Intervention,; Latino, farm worker; randomized controlled intervention
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2 | interventions — Behavior Therapy; Diet

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral intervention (Experimental): Behavioral intervention consisting of 10 educational sessions promoting healthy diet and increased physical activity.
  Interventions: Behavioral: Behavioral Intervention
- Control (Active Comparator): Control arm received no behavioral intervention
  Interventions: Behavioral: Behavioral Intervention

INTERVENTIONS:
Behavioral: Behavioral Intervention — Intervention participants attended up to 10 educational sessions teaching them about diabetes, and modifiable lifestyle factors (behaviors) to reduce the risk of diabetes by controlling weight. Sessions were conducted by Promotoras using culturally sensitive and appropriate materials and themes. Group activities and support were also emphasized. The control participants like the intervention were measured and interviewed before and again after the intervention sessions, but received no educational instruction or materials.
  Other Names: Healthy Lifestyle intervention; Diet and Physical Activity intervention

SUMMARY:
This is a study to assess the effectiveness of a culturally appropriate behavioral intervention to reduce obesity levels and ultimately the risk of developing diabetes type II in immigrant Latino farm workers. Workers enrolled in a 2:1 ratio by random allocation into an intervention or control arm of the study. The intervention participants received weekly classes for 10 weeks with education on diabetes, diet and physical activity and practical exercises. Both control and intervention were measured for weight, waist circumference, fasting blood glucose and interviewed before and after the study intervention. The main hypothesis was that intervention, but not control participants, would experience reduction in body measurements after the intervention.

DETAILED DESCRIPTION:
A more detailed description is not desired as noted above.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 -60
* BMI between 20 -38
* Willing to attend 10 weekly education sessions
* Able to speak and understand Spanish
* Have medical insurance

Exclusion Criteria:

* Fasting blood glucose about 126mg/dL unless physician attests fit to participate
* Pregnancy or trying to conceive, or breastfeeding
* Diabetic
* On therapeutic diets
* On medications that affect weight
* If spouse / cohabitant already in the study
* Not a farm worker working for the Reiter Affiliated Companies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 254 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change in BMI | Before intervention and after (12-14 weeks after first assessment)
  Weight and Height assessed for both control and intervention participants before intervention program and then assessed 2-3 weeks after the intervention period completed.

SECONDARY OUTCOMES:
Change in Waist Circumference | Measured before and after intervention (12 - 13 weeks after first assessment
  Waist circumference measured in both control and intervention participants using a standard protocol. Conducted before intervention started and again 2-3 weeks after the intervention sessions finished.

OTHER OUTCOMES:
Change in fasting blood glucose | Measured before intervention and after (12-13 weeks after first assessment)
  Fasting blood glucose was a voluntary assessment and therefore not conducted in all participants. Blood glucose was assessed from a middle digit using a sterile lancet and Accu-Check Advantage Blood Glucose Meter. It was assessed before the start of the intervention and after completion in both controls and intervention participants.

CONTACTS AND LOCATIONS:
Overall Officials: Marc B Schenker, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - Reiter Affiliated Companies, Oxnard, California
  - Reiter Affiliated Companies, Watsonville, California

REFERENCES:
- [Derived] Mitchell DC, Andrews T, Schenker MB. Pasos Saludables: A Pilot Randomized Intervention Study to Reduce Obesity in an Immigrant Farmworker Population. J Occup Environ Med. 2015 Oct;57(10):1039-46. doi: 10.1097/JOM.0000000000000535. PMID 26461858